CLINICAL TRIAL: NCT01721434
Title: Effects of Levosimendan on Diaphragm Function in Mechanically Ventilated Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Nijmegen (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Principal Investigator, Leo Heunks, MD, PhD, University Medical Center Nijmegen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Levo2
Record Dates: First submitted 2012-09-21; First posted 2012-11-05 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Muscle Weakness Conditions; Weaning Failure
Keywords: levosimendan; diaphragm function; mechanically ventilated patients; neuro-mechanical efficiency
MeSH Terms: interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levosimendan (Experimental): Levosimendan 0.2 ug/kg/min intravenous for a single 7 hours.
  Interventions: Drug: Levosimendan
- Placebo (Placebo Comparator): Similar coloured placebo intravenous for a single 7 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levosimendan
  Other Names: Simdax
  Arms: Levosimendan
Drug: Placebo — Similar coloured placebo
  Arms: Placebo

SUMMARY:
Levosimendan is a relatively new drug that improves cardiac contractility in patients with heart failure. Its main mechanism of action is enhanced binding of calcium to the myocardial contractile proteins. Recent data from our lab showed that levosimendan improves contractility of human diaphragm in vitro (muscle fibers from COPD patient diaphragm) and in vivo (healthy subjects). Accordingly, levosimendan may appear of value in the treatment of disorders associated with impaired respiratory muscle function, such as mechanically ventilated patients.We hypothesize that levosimendan could improve respiratory muscle function in mechanically ventilated patients commencing a CPAP trial.

ELIGIBILITY:
Inclusion Criteria:

* mechanical ventilation > 3 days
* informed consent
* able to sustain a CPAP trial for 30 minutes
* PaO2/FiO2 ratio > 200 mmHg
* ventilatory settings: positive end expiratory pressure <= 10 cmH2O, pressure support <= 10 cmH2O

Exclusion Criteria:

* pre-existent muscle disease (congenital or acquired) or diseases/disorders known to be associated with myopathy including auto-immune diseases
* pre-existent cardiac disease (based on history, electrocardiography and transthoracic echocardiography)
* upper airway/esophageal pathology (i.e. recent surgery, esophageal varices, diaphragmatic hernia)
* phrenic nerve lesions
* pregnancy, breast feeding
* severe renal failure (serum creatinine > 150 umol/L)
* severe hepatic failure
* recent (within 5 days) nasal bleeding
* systolic blood pressure < 120 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Neuro-mechanical efficiency of the diaphragm | Artefact-free periode in the last 10 minutes of each CPAP trial
  The primary outcome measure is the neuro-mechanical efficiency(i.e. the ratio of diaphragm electrical activity and transdiaphragmatic pressure) of the diaphragm during a continuous positive airway pressure (CPAP) trial.

SECONDARY OUTCOMES:
Neuro-ventilatory efficiency of the diaphragm | Artefact-free periode in the last 10 minutes of each CPAP trial
  A secondary outcome measure is the neuro-ventilatory efficiency (i.e. the ratio of diaphragm electrical activity and tidal volume) during a continuous positive airway pressure (CPAP) trial.
Oxygen consumption (VO2) | Artefact-free periode in the last 10 minutes of each CPAP trial
  A secondary outcome measure is the oxygen consumption during a continuous positive airway pressure (CPAP) trial.
Partial pressure of oxygen in arterial blood (PaO2) | Last minute of the 30 minute CPAP trial
  A secondary outcome measure is the PaO2 at the end of a continuous positive airway pressure (CPAP) trial.
Accessory respiratory muscle activity | Measured during a one hour protocol after the second CPAP trial.
  To determine the effects of levosimendan on accessory respiratory muscle function, ventilator settings are adapted after the last CPAP-trial.
Carbon dioxide production (VCO2) | Artefact-free periode in the last 10 minutes of each CPAP trial
  A secondary outcome measure is the carbon dioxide production during a continuous positive airway pressure (CPAP) trial.
Partial pressure of carbon dioxide in arterial blood (PaCO2) | Last minute of the 30 minute CPAP trial
  A secondary outcome measure is the PaCO2 at the and of a continuous positive airway pressure (CPAP) trial.

CONTACTS AND LOCATIONS:
Overall Officials: Leo Heunks, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands